CLINICAL TRIAL: NCT01922830
Title: Probiotics and Microbiota in Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director, r&d division, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-13-OS-196-CTIL
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: NAFLD
Keywords: Sleeve Gastrectomy; NAFLD; gut microbiot; Bariatric surgery
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bio-25 (Supherb) (Experimental): Bio-25 (Supherb) once daily (2 capsules -50 billion bacteria) for 6 months (or 4 weeks for healthy participants).
  The Bio-25 (Supherb) is a probiotic supplement consisting of 11 different species of patented probiotic bacteria and over 25 billion active bacteria in each capsule. The bacteria in the formula are patented bacteria that have undergone drying, freezing, and double coating which ensures their survival under stomach acidity conditions and their enrooting in the intestines.
  Interventions: Dietary Supplement: Bio-25 (Supherb)
- Placebo (Placebo Comparator): Identical placebo once daily (2 capsules) for 6 months (or 4 weeks for healthy participants).
  The placebo supplementation is identical-looking to the Bio-25 supplement.
  Interventions: Dietary Supplement: Placebo (for Bio-25, Supherb)

INTERVENTIONS:
Dietary Supplement: Bio-25 (Supherb) — The Bio-25 (Supherb) is a probiotic supplement consisting of 11 different species of patented probiotic bacteria and over 25 billion active bacteria in each capsule. The bacteria in the formula are patented bacteria that have undergone drying, freezing, and double coating which ensures their survival under stomach acidity conditions and their enrooting in the intestines.
  Arms: Bio-25 (Supherb)
Dietary Supplement: Placebo (for Bio-25, Supherb) — A pill manufactured to mimic Bio-25 (Supherb) pill
  Arms: Placebo

SUMMARY:
This study is a randomized clinical trial with 6 months probiotic supplement vs. placebo treatment and 6 month follow up on 100 NAFLD patients that will undergo sleeve gastrectomy surgery. Measurements will be conducted at: baseline, M3 (3 months after treatment initiation), M6 and M12 and will include: abdominal US, Fibroscan, biochemical tests, anthropometric measurements, glucose breath test for bacterial overgrowth, fecal samples and questionnaires for demographic details, quality of life, food intake, food tolerance and habitual physical activity. 20 subjects will undergo an additional liver-MRI test at baseline and M6.

Additionally, 30 healthy participants will consume probiotic supplement vs. placebo for 28 days and will undergo gastroscopy and colonoscopy before and during consumption.

DETAILED DESCRIPTION:
Background:

Bariatric surgery is an effective and increasingly common treatment for obesity and obesity-related comorbidities. Among patients undergoing bariatric surgery, as many as 96% have NAFLD (Nonalcoholic fatty liver disease) and up to 25% have NASH (Nonalcoholic steatohepatitis). Intestinal microbiota has been shown to play pivotal roles in host mammalian developmental, immune and metabolic functions. Alterations in the gut microbiome, or 'dysbiosis' has been recently linked to the pathogenesis of metabolic disease including obesity, insulin resistance, atherosclerosis and liver diseases. Recent studies show that modulation of gut microbiota may represent a novel way to treat or prevent NAFLD and its progression. Bariatric surgery is associated with major modifications in microbiota composition, quantity and function. Potential mediators to the gut microbiota are probiotics which are considered to be a safe therapy since its microorganisms composition is found naturally in human microflora. Clinical research has shown that probiotic supplementation can induce physiological changes in the intestinal flora (e.g., via the secretion of endogenic antibiotics and other defensins). Moreover, It was shown that probiotic bacteria are assimilated in the gut mucosa, thus replacing and changing the natural bacterial line-up. The biopsies taken in the healthy section of the study will help us evaluate all the above changes, after 4 weeks of probiotic intervention.

To date, there is lack of evidence on the use of probiotics in bariatric surgeries with just 1 randomizes clinical trial in Roux-en-Y gastric bypass surgery patients.

Aims:

To evaluate the effect of 6 months probiotic supplement vs. placebo on clinical and metabolic parameters in patients with NAFLD undergoing sleeve gastrectomy surgery.

Working hypothesis: Modulation of gut microbiota with probiotic will have a beneficial effect on clinical and metabolic parameters in sleeve gastrectomy patients with NAFLD.

To evaluate the effect of 4 weeks probiotic supplement vs. placebo on microbiome composition and function in healthy volunteers.

Methods:

A randomized double blind clinical trial with 6 months treatment and 6 months follow up including 2 treatment arms: probiotic and placebo. One hundred NAFLD patients who will undergo sleeve gastrectomy surgery through the bariatric surgery clinic at the Tel Aviv Assuta medical center will be enrolled during 2013-2016. Baseline and follow up evaluation will be performed at the Tel-Aviv Sourasky Medical center and will include: abdominal US (hepato-renal index-HRI), Fibroscan, biochemical tests, anthropometric measurements, glucose breath test for bacterial overgrowth (BO). Fecal samples will be collected and analyzed for gut microbiota utilizing 'state of the art' molecular methods. All patients will fill out validated questionnaires of demographic details, quality of life, food intake, food tolerance and habitual physical activity. Measurements will be conducted at: baseline, M3 (3 months after treatment initiation), M6 and M12. 20 subjects will undergo an additional liver-MRI test at baseline and M6.

Importance of the study: Almost all morbid obese patients have NAFLD and up to 25% have NASH, leading to major hepatic and extra-hepatic complications. Only limited data are available concerning gut microbiota composition after bariatric surgery and its association with weight reduction, metabolic and hepatic parameters. Moreover, there are no clinical trials on the role of probiotics administration following sleeve gastrectomy bariatric surgery on hepatic parameters. Probiotic supplement after bariatric surgery may improve the therapeutic effect of the surgery on hepatic steatosis and may improve also biochemical tests of vitamins (e.g. B12), inflammatory mediators (e.g. endotoxin levels) and metabolic parameters, reduce bacterial overgrowth and enhance weight loss. The study would help in developing new treatment approaches and will contribute to the understanding of the mechanisms underlying the hepatic, metabolic and inflammatory consequences of bariatric surgery.

Probiotic supplement vs. placebo will be given to 30 healthy participants. participants will undergo gastroscopy (upper GI endoscopy) + colonoscopy (lower GI endoscopy) before the probiotics intervention and after 3 to 4 weeks of probiotic intervention. During the procedure, biopsies will be taken from different segments of the GI tract. The study samples will be frozen performing the microbial tests. In addition, participants will collect fecal samples. In this section, participants will be followed-up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-65 years old
* BMI > 40 kg/m² or BMI > 35 kg/m² with comorbidities (See Appendix 1 for the Ministry of health indications for bariatric surgeries) that got the bariatric commission approval of Assuta private hospitals to undergo sleeve gastrectomy surgery
* Willingness to take a probiotic/placebo supplement once a day for 6 months
* Ultrasound diagnosed NAFLD patients
* Reading and speaking Hebrew

Healthy volunteers:

* Subjects 18-65 years old
* Healthy subjects

Exclusion Criteria:

* Subject with mental illness or cognitive deterioration
* Use of probiotic/antibiotic 3 mounts before surgery
* Use of other antibiotic for more than 1 week during the study
* Drug addiction
* Excessive alcohol consumption (≥ 30 g/day in men or ≥ 20 g/day in women)
* Treatment with drugs known to cause hepatic steatosis or elevation of liver enzymes (e.g. Corticosteroids, HAART, Amiodarone, high dose estrogens) (see Appendix 2)
* Treatment with drugs or supplements that may improve hepatic steatosis or liver enzymes (Vitamin E, Milk thistle, ω-3 fatty acid, Ursodeoxycholic acid) 3 months prior to the initiation of the study
* Other causes of chronic liver disease ( e.g. viral hepatitis: HBV/HCV +, autoimmune hepatitis, Hemochromatosis, Wilson's disease)
* Diabetic patients who are treated with antidiabetic medications, except diabetic patients who are treated for at least 6 months exclusively with Metformin at a stable dose
* Subjects who began a new lipid reduction medications less than 6 months prior to the initiation of the study
* Subjects with chronic conditions that could interfere with our study: active cancer, organ transplant subjects, advanced kidney or liver disease, inflammatory bowel disease and other systemic inflammatory conditions
* Bariatric surgery in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Hepato-Renal Index (HRI) method by abdominal US | 36 months
  US will be performed at pretrial, 6 ,12 , 36 months after the surgery. .Fatty liver will be diagnosed by abdominal US using standardized criteria. HRI, a validated quantitative measure, will be calculated on the basis of the ratio between the echogenicity of the liver and that of the right kidney cortex using histogram echo intensity.

SECONDARY OUTCOMES:
Liver fibrosis - by Fibroscan (transient elastography) | 36 months
  The liver stiffness will be measured by Fibroscan (using XL probe) and will be performed at pretrial, 6 and 12 month after the surgery. The liver stiffness is measured by Fibroscan in a volume of approximates 1 cm wide and 4 cm long cylinder, representing 1/500 of liver tissue (100 times greater than a biopsy sample). The results of the Fibroscan test are expressed in KiloPascals (kPa). The Fibroscan XL probe reduces Fibroscan failure and facilitates reliable liver stiffness measurement in obese patients compared with the common M probe.
Anthropometric measurements | 36 months
  Measurements of anthropometry will be performed following a uniform protocol at pretrial, 3, 6 and 12 month after the surgery. Height, weight, WC (Waist circumference) will be measured. BMI and %EWL will be calculated. "Tanita" will be used for body composition analysis (%fat mass, fat mass and fat free mass) and will be performed at pretrial and 6 month after the surgery.
Biochemical fasting blood tests | 36 months
  Patients will undergo biochemical tests at pretrial, 3, 6 ,12, 36 months after the surgery. All blood samples will be drawn at the morning after a fast of at least 12 hours. Serological tests that will be taken: lipid profile, inflammatory factors (CRP, TNF-α, IL6, IL10, TGF- β), adipocytokines (leptin, adiponectin), endotoxin (Lipopolysacchride), hepatocyte apoptosis markers (CK-18, sFas), glucose, HbA1C, total bilirubin, liver enzymes, TSH, insulin, vitamin B1, vitamin B12, vitamin D, Iron, ferritin, folic acid. HOMA will be calculated as: serum insulin (μIU/ml) x plasma glucose (mmol/l)/22.5. HOMA index ≥2.77 is considered to be diagnostic for insulin resistance.
The fecal microbiota composition | 6 years
  Fecal samples will be taken at pretrial and 6 month after the surgery. Fecal samples will be obtained in the morning before breakfast. The stools will be self-collected in sterile boxes that will be given to the participants in advance and will be stored at -800C degrees until further analysis. DNA will be extract from feces for detecting microbiota diversion. Philogenetic analysis will be performed using pyrosequencing and multiplexing of bacterial 16S rRNA segments. Samples from several randomly selected individuals will be used for shotgutn metagenomic sequencing.
Quality of life (QoL) | 36 months
  Patients will fill out a self-reported QoL questionnaire at pretrial, 3, 6 , 12, 36 month after the surgery. The SF-12 (a shorter version of the SF-36) is a QoL questionnaire. The SF-12 yields 2 summary scores: physical component summary (PCS) and mental component summary (MCS). The SF-12 have been translated and validated in many languages (including Hebrew) and were found valid and reliable among the general population. Higher scores on the PCS and MCS indicate better health.
Food tolerance after bariatric surgery | 36 months
  Patients will fill out a self-reported questionnaire for quick assessment of food tolerance after bariatric surgery at pretrial, 3, 6 and 12 month after the surgery. To evaluate food tolerance we will use this questionnaire which was previously described by Suter et al. This questionnaire is simple to fill out, reliable, and useful both in following up individuals after bariatric surgery and in comparing results after different procedures as part of the evaluation of QoL . The score for this questionnaire is divided into 3 parts: Patient's satisfaction of their food intake, food tolerance (for 8 different types of food) and the frequency of vomiting/regurgitation.
Liver MRI | 6 months
  20 subjects will undergo an additional liver-MRI test at baseline and M6.
Hand grip | 36 months
  For hand dynamometer a standard chair with a straight back without arm rests is needed. The participant sits in a chair with his/her feet flat on the floor and his/her knees at 90-degree angle. The arm being tested should be at a 90-degree angle, next to but not touching his body. The tester demonstrates the test and then the participant does a practice trial on the dominant and then the non-dominant hand. After the practice trial the examiner will put the dynamometer in the participants dominant hand and with saying "Go" the subject will squeeze his hand as hard as possible for 3-4 seconds till examiner says 'stop'. The maximum reading will be recorded. The participant will then perform the test once more on the non-dominant hand. Measurement will be recorded. A 2 trials / hand (15 seconds rest between trails) will be performed in alternate fashion and best score (in kg) will be recorded.
Microbiome composition and function | 6 years
  Gastrointestinal tract biopsies, fecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Oren Shibolet, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Sherf-Dagan S, Zelber-Sagi S, Buch A, Bar N, Webb M, Sakran N, Raziel A, Goitein D, Keidar A, Shibolet O. Prospective Longitudinal Trends in Body Composition and Clinical Outcomes 3 Years Following Sleeve Gastrectomy. Obes Surg. 2019 Dec;29(12):3833-3841. doi: 10.1007/s11695-019-04057-2. PMID 31301031
- [Derived] Shenhar-Tsarfaty S, Sherf-Dagan S, Berman G, Webb M, Raziel A, Keidar A, Goitein D, Sakran N, Zwang E, Shapira I, Zeltser D, Berliner S, Rogowski O, Shibolet O, Zelber-Sagi S. Obesity-related acetylcholinesterase elevation is reversed following laparoscopic sleeve gastrectomy. Int J Obes (Lond). 2019 Feb;43(2):297-305. doi: 10.1038/s41366-018-0014-4. Epub 2018 Feb 3. PMID 29491490
- [Derived] Sherf Dagan S, Zelber-Sagi S, Webb M, Keidar A, Raziel A, Sakran N, Goitein D, Shibolet O. Nutritional Status Prior to Laparoscopic Sleeve Gastrectomy Surgery. Obes Surg. 2016 Sep;26(9):2119-2126. doi: 10.1007/s11695-016-2064-9. PMID 26797718